CLINICAL TRIAL: NCT04052152
Title: Anlotinib Hydrochloride Capsules Combined With Sintilimab Injection in the Treatment of Advanced Hepatocellular Carcinoma (HCC) Open, Single Arm, Exploratory Clinical Trial
Brief Title: Anlotinib Hydrochloride Combined With Sintilimab Injection in the Treatment of Advanced Hepatocellular Carcinoma (HCC)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KEEP-G 04
Record Dates: First submitted 2019-07-16; First posted 2019-08-09 (Actual); Last update posted 2019-08-09 (Actual); Status verified 2019-07

CONDITIONS: Advanced Hepatocellular Carcinoma
Keywords: HCC; Antiangiogenic agents combined with PD-1 antibody
MeSH Terms: interventions — anlotinib; sintilimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Group A (Experimental): Patients in the study group will receive the following treatment:
  21 days as a treatment cycle, Anlotinib 12mg/day(D1-D14 ) and Sintilimab injection 200mg Q3W (D1). Sintilimab injection will be administered until disease progressioncor un-tolerable toxicity. Anlotinib will be administered until disease progression. If anlotinib is not tolerated, the dose can be reduced to 10mg or 8mg ,until un-tolerable toxicity again
  Interventions: Drug: Anlotinib and Sintilimab injection

INTERVENTIONS:
Drug: Anlotinib and Sintilimab injection — Patients will be treated with Anlotinib and Sintilimab injection

SUMMARY:
This is a single-arm, open-label and exploratory clinical study of Anlotinib Hydrochloride Capsules combined with Sintilimab injection in the treatment of advanced Hepatocellular Carcinoma (HCC).

In oder to observe and evaluate the efficacy and safety of Anlotinib Hydrochloride Capsules combined with Sintilimab injection. Subjects with pathological confirmed Hepatocellular Carcinoma will be enrolled.

21 days as a treatment cycle, Anlotinib 12mg/day(D1-D14 ) and Sintilimab injection 200mg Q3W (D1). Sintilimab injection will be administered until disease progressioncor un-tolerable toxicity. Anlotinib will be administered until disease progression. If anlotinib is not tolerated, the dose can be reduced to 10mg or 8mg ,until un-tolerable toxicity again.

DETAILED DESCRIPTION:
This is a single-arm, open-label and exploratory clinical study of Anlotinib Hydrochloride Capsules combined with Sintilimab injection in the treatment of advanced Hepatocellular Carcinoma (HCC).In oder to observe and evaluate the efficacy and safety of Anlotinib Hydrochloride Capsules combined with Sintilimab injection.subjects with pathological confirmed Hepatocellular Carcinoma will be enrolled.21 days as a treatment cycle, Anlotinib 12mg/day(D1-D14 ) and Sintilimab injection 200mg Q3W (D1). Sintilimab injection will be administered until disease progressioncor un-tolerable toxicity. Anlotinib will be administered until disease progression. If anlotinib is not tolerated, the dose can be reduced to 10mg or 8mg ,until un-tolerable toxicity again.

ELIGIBILITY:
Inclusion criteria:

1. At least one measurable lesion (the length of spiral CT scan (> 10mm) meets the requirements of RESCIST 1.1) is found in patients with HCC confirmed by histopathology or cytology or who meet the clinical diagnostic criteria.
2. Inability or unwillingness to undergo surgery and transcatheter hepatic artery interventional therapy; if interventional therapy, radiotherapy or surgery has been accepted, it must be more than 4 weeks, and adverse reactions or wounds have fully recovered.
3. No treatment with sorafenib or other systemic treatment was received. Patients who have used interventional chemotherapeutic drugs during interventional therapy may be enrolled in the group.
4. Child-Pugh liver function rating: grade A or B; BCLC stage B or C.
5. ECOG 0-1
6. The life expectancy is more than 12 weeks.
7. The main organs are functioning normally.
8. Subjects volunteered to join the study, signed informed consent, good compliance, with follow-up.

Exclusion Criteria:

1. Hepatobiliary and mixed cell carcinomas and fiberboard cell carcinomas are known; other malignant tumors (except cured cutaneous basal cell carcinomas and cervical carcinoma in situ) have been reported in the past or at the same time.
2. Pregnant or lactating women.
3. Patients with hypertension who could not be well controlled by antihypertensive drugs (systolic blood pressure > 150 mmHg, diastolic blood pressure > 100 mmHg), patients with myocardial ischemia or myocardial infarction above grade II, arrhythmias with poor control (including QTC interval > 450 ms) and cardiac insufficiency of grade III-IV according to NYHA standard.
4. Inability to swallow, chronic diarrhea and intestinal obstruction significantly affect drug use and absorption.
5. There are clear concerns about gastrointestinal bleeding (such as local active ulcer lesions, fecal occult blood ++) or more), and there is a history of gastrointestinal bleeding within 6 months.
6. Coagulation dysfunction (PT > 16 s, APTT > 43 s, TT > 21 s, Fbg < 2 g/L), with bleeding tendency or undergoing thrombolysis or anticoagulation therapy.
7. Have a history of mental illness or psychotropic drug abuse.
8. Peritoneal effusion with clinical symptoms requires therapeutic abdominal puncture or drainage. Or patients with hepatic encephalopathy as well as with liver transplantation.
9. Patients with cancer thrombus involving the main portal vein or inferior vena cava.
10. Patients with Infectious pneumonia, non-infectious pneumonia, interstitial pneumonia and other disease requiring corticosteroids.
11. A history of chronic autoimmune diseases, such as systemic lupus erythematosus.
12. Patients with a history of inflammatory bowel diseases such as ulcerative enteritis and crohn's disease. Or patients with a history of inflammatory chronic diarrheal diseases such as irritable bowel syndrome.
13. Patients with a history of sarcoidosis or tuberculosis.
14. Patients with active hepatitis b, c and HIV infection; HBVER who could controll HBV DNA<500 copy/ml after antiviral treatment is allowed to be included.
15. Patients who are allergic to components of Sintilimab injection and anlotinib preparations, or have a history of severe allergic reactions to other monoclonal antibodies.
16. Having a history of psychotropic substance abuse and being unable to quit or having a mental disorder.
17. Patients with a history of immunodeficiency, or other acquired congenital immunodeficiency diseases, or a history of organ transplantation and hematopoietic stem cell transplantation.
18. First dose immunosuppressive drugs used in the first 4 weeks, not including the nasal spray, inhalation, or other ways of topical corticosteroids or physiological doses of systemic corticosteroids (no more than 10 mg/day prednisone or other equivalent dose glucocorticoids). But temporary use of glucocorticoids is permitted for the treatment of dyspnea symptoms of asthma, chronic obstructive pulmonary disease and other diseases.
19. Systemic immunostimulant therapy was administered within 4 weeks prior to first administration or planned during the study period. Or systemic immunostimulant therapy was received within 4 weeks.
20. According to the researchers' judgment, there are serious concomitant diseases that endanger patient safety or prevent patients from completing the study.
21. Drug combinations that have an effect on the metabolism of CYP3A.
22. Urinary protein 2+ or 24-hour urinary protein >1g.
23. Central nervous system metastasis has occurred.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-06-10 (Actual); Primary Completion 2019-12-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 18 months
  the best Objective Response Rate
Adverse reaction rate | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 18 months
  Observe all the participants in any adverse events occurred during the period of clinical research, including clinical symptoms and signs of life, an abnormal in laboratory tests, record its clinical characteristics, severity, occurrence time, duration, treatment and prognosis, and determine its and the correlation between test drugs. NCI-CTC AE 5.0 standard was used to evaluate drug safety.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 18 months
  Progression Free Survival
Duration of Response (DOR) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 18 months
  Duration of Response
Disease Control Rate (DCR) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 18 months
  the Rate of Disease Control
Overall survival (OS) | From date of randomization until the date of patient died, assessed up to 24 months
  Overall Survival

CONTACTS AND LOCATIONS:
Overall Officials: Yongqian Shu, PhD, Principal Investigator — JANGSU PROVINCE HOSPITAL
Locations (1):
- Jiangsu Province Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen X, Li W, Wu X, Zhao F, Wang D, Wu H, Gu Y, Li X, Qian X, Hu J, Li C, Xia Y, Rao J, Dai X, Shao Q, Tang J, Li X, Shu Y. Safety and Efficacy of Sintilimab and Anlotinib as First Line Treatment for Advanced Hepatocellular Carcinoma (KEEP-G04): A Single-Arm Phase 2 Study. Front Oncol. 2022 May 31;12:909035. doi: 10.3389/fonc.2022.909035. eCollection 2022. PMID 35712486